CLINICAL TRIAL: NCT07284914
Title: Community Interventions for Tackling Antimicrobial Resistance in Ghana
Acronym: CITAR-Ghana
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: University of Ghana (Other)
Responsible Party: Principal Investigator, Yubraj Acharya, Ph.D., Associate Professor, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: STUDY00026602; 102725 (Other Grant/Funding Number: Merck and Company, Inc.)
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Upper Resp Tract Infection
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: Community pharmacies will be randomized into 3 arms (control, Individualized Feedback, and Legal Reminder). Pharmacies in each arm will be visited by standardized patients under 4 scenarios (low demand-young patient; low demand-old patient, normal demand-young patient, normal demand-old patient).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): No intervention
- Individualized Feedback (Experimental): Pharmacies receive customized feedback on their antibiotics dispensing behavior.
  Interventions: Behavioral: Individualized Feedback
- Legal Reminder (Experimental): Pharmacies receive letter from the authorities in Ghana emphasizing that providing antibiotics without a physician prescription is against the law.
  Interventions: Behavioral: Legal Reminder

INTERVENTIONS:
Behavioral: Individualized Feedback — We use information from the baseline visits (e.g., on whether they give antibiotics without a prescription and the time they spend with patients) to provide customized feedback to the pharmacies.
  Arms: Individualized Feedback
Behavioral: Legal Reminder — We provide a letter from the authorities in Ghana emphasizing that providing antibiotics without a physician prescription is against the law.
  Arms: Legal Reminder

SUMMARY:
This research project aims to test the effect of two interventions targeted to community pharmacies in the Greater Accra region, Ghana, on antibiotics dispensing rates. The general goal is to inform the design of future policies to address the rising threat of antimicrobial resistance.

DETAILED DESCRIPTION:
Interventions that discourage community pharmacies from providing antibiotics without proper diagnosis and a physician's prescription are critically needed in low- and middle-income countries in order to address the rising threat of antimicrobial resistance. In this study, we will test the effect of two interventions targeted to community pharmacies in the Greater Accra region of Ghana. We will conduct a baseline survey, followed by visits by standardized patients (SPs). We will then implement the interventions (described below) and assess the outcomes again using SPs.

The study has 4 key objectives:

Objective 1. Assess the effect of two behavioral interventions targeted to community pharmacies on antibiotics dispensing rates. We randomly assign 285 pharmacies in Greater Accra 1:1:1 into one of three arms: 1) Control, 2) Individualized Feedback, and 3) Legal Reminder. In the Individualized Feedback arm, we use information from the first visits to provide customized feedback to the pharmacies. In the Legal Reminder arm, we provide a letter from the Ghana authorities emphasizing that providing antibiotics without a physician prescription is against the law.

Objective 2. Assess the extent of know-do gap in antibiotics dispensing behavior among community pharmacies. We compare self-reported data from a baseline survey and the one obtained from SP visits to assess the gap between what the pharmacies know and what they do in practice.

Objective 3. Examine the effect of reduced pressure from patients for antibiotics on pharmacies' dispensing behavior. The two demand variations we will test are the following: 1) Patient asks for a medicine (normal demand pressure), 2) Patient explicitly says that they would prefer not to take antibiotics and mention that they do not have a physician prescription and that their condition appears to be viral (reduced demand pressure).

Objective 4. Assess differential effects of the two interventions and reduced demand pressure across patient's age.

ELIGIBILITY:
Inclusion Criteria for community pharmacies:

* Operating within the Greater Accra region of Ghana
* Registered with Ghana Pharmacy Council
* "Stand-alone", i.e., not affiliated or next to a hospital

Exclusion Criteria:

* Operating only outside the Greater Accra region of Ghana
* Not registered with Ghana Pharmacy Council
* Hospital pharmacy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 285 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Non-prescription antibiotics dispensing rate | From baseline (1st SP visit) to the final SP visit (visit 5), lasting approximately 5 months.
  Whether the pharmacy dispenses antibiotics without prescription in scenarios not requiring them

SECONDARY OUTCOMES:
Watch or reserve antibiotics | From baseline (1st SP visit) to the final SP visit (visit 5), lasting approximately 5 months.
  Whether the dispensed antibiotics fall into the Watch or Reserve category in the WHO AWaRE classification.
Out-of-pocket costs to patients | From baseline (1st SP visit) to the final SP visit (visit 5), lasting approximately 5 months.
  Amount patients spend out-of-pocket on medications including antibiotics.
Referral to a physician | From baseline (1st SP visit) to the final SP visit (visit 5), lasting approximately 5 months.
  Whether the pharmacist recommends the patient to see a doctor before antibiotics can be dispensed.
History taking | From baseline (1st SP visit) to the final SP visit (visit 5), lasting approximately 5 months.
  Number of questions asked by the pharmacist based on a pre-specified checklist of appropriate history taking behavior
Interaction time | From baseline (1st SP visit) to the final SP visit (visit 5), lasting approximately 5 months.
  Amount of time the pharmacist spends on the patient before giving medicine.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ghana, Regional Institute for Population Studies, Legon, Ghana

IPD SHARING:
Plan to Share IPD: No